CLINICAL TRIAL: NCT00365105
Title: Randomized Phase III Trial to Evaluate Radiopharmaceuticals and Zoledronic Acid in the Palliation of Osteoblastic Metastases From Lung, Breast, and Prostate Cancer
Brief Title: Zoledronate, Vitamin D, and Calcium With or Without Strontium 89 or Samarium 153 in Preventing or Delaying Bone Problems in Patients With Bone Metastases From Prostate Cancer, Lung Cancer, or Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RTOG 0517; CDR0000491233; NCI-2009-00727 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Results first posted 2014-11-10 (Estimated); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer; Lung Cancer; Metastatic Cancer; Pain; Prostate Cancer
Keywords: pain; bone metastases; extensive stage small cell lung cancer; recurrent breast cancer; stage IV breast cancer; recurrent non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Neoplasm Metastasis; Pain; Prostatic Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Calcium; Vitamin D; Zoledronic Acid; Samarium-153; strontium chloride; Strontium-89

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zoledronic acid (Active Comparator): Zoledronic acid, vitamin D and calcium supplements.
  Interventions: Dietary Supplement: Calcium; Dietary Supplement: Vitamin D; Drug: zoledronic acid
- Zoledronic acid + Radiopharmaceuticals (Experimental): Zoledronic acid, vitamin D and calcium supplements, plus Sr-89 or Sm-153.
  Interventions: Dietary Supplement: Calcium; Drug: zoledronic acid; Drug: Sm-153; Radiation: Sr-89

INTERVENTIONS:
Dietary Supplement: Calcium — At least 500 mg of calcium (1 pill) by mouth daily until the study doctor thinks it is in their best interest to stop.
Dietary Supplement: Vitamin D — 400 IU of vitamin D (1 pill) by mouth daily until the study doctor thinks it is in their best interest to stop.
  Arms: Zoledronic acid
Drug: zoledronic acid — 4 mg of Zoledronic acid intravenously once a month until the study doctor thinks it is in their best interest to stop.
  Other Names: Zometa
Drug: Sm-153 — Single dose intravenously 1 mCi/kg body weight.
  Other Names: Samarium-153
  Arms: Zoledronic acid + Radiopharmaceuticals
Radiation: Sr-89 — Single dose intravenously 4 mCi.
  Other Names: Strontium-89
  Arms: Zoledronic acid + Radiopharmaceuticals

SUMMARY:
RATIONALE: Zoledronate, vitamin D and calcium may prevent or delay bone pain and other symptoms caused by bone metastases. It is not yet known whether giving zoledronate together with vitamin D and calcium is more effective with or without strontium 89 or samarium 153 in treating patients with bone metastases from prostate cancer, lung cancer, or breast cancer.

PURPOSE: This randomized phase III trial is studying zoledronate, vitamin D, and calcium to see how well they work compared to zoledronate, vitamin D, calcium, and either strontium 89 or samarium 153 in preventing or delaying bone problems in patients with bone metastases from prostate cancer, lung cancer, or breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of zoledronate, vitamin D, and calcium with or without strontium chloride Sr 89 or samarium Sm 153 lexidronam pentasodium, in terms of preventing or delaying the time to development of malignant skeletal-related events (SREs) (defined as a pathological bone fracture, spinal cord compression, surgery to bone, or radiation to bone) in patients with bone metastases secondary to prostate, lung, or breast cancer.

Secondary

* Compare the rate of SREs at 1 year in patients treated with these regimens.
* Compare overall survival of patients treated with these regimens.
* Compare quality of life of patients treated with these regimens.
* Compare the effect of these regimens on pain control in these patients.
* Evaluate resource utilization and cost effectiveness of these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to primary disease site (prostate vs breast vs lung) and number of bone metastases (≤ 2 vs > 2). Patients are randomized to 1 of 2 treatment arms.

Quality of life and pain are assessed at baseline and then at 1, 3, 6, and 12 months from start of protocol treatment.

After completion of study treatment, patients are followed every 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven diagnosis of solid tumor malignancy of lung, breast, or prostate prior to registration;
2. Appropriate diagnosis for protocol entry, based upon the following minimum diagnostic workup:

   2.1 History/physical examination within 8 weeks prior to registration; 2.2 Bone scan within 4 weeks prior to registration; bone metastases must be visible on the scan. Other scanning modalities, such as magnetic resonance imaging (MRI), positron emission tomography (PET) 2.3 Dental evaluation according to the dental exam checklist (carried out by the investigator, the investigator's designee, or by a qualified dental professional [dental hygienist or dentist]), including history of dental surgery (e.g., extraction or implant) within 8 weeks prior to registration and recorded on the dental exam checklist; Note: If the patient has received prior oral bisphosphonate therapy and has had a prior dental evaluation within 8 weeks of registration, the evaluation should not be repeated.

   2.4 Complete blood count (CBC)/differential within 2 weeks prior to registration, with adequate bone marrow function defined as follows:
   * White blood cell count (WBC) ≥ 2400 cells/mm^3;
   * Absolute neutrophil count (ANC) ≥ 1,800 cells/mm3;
   * Platelets ≥ 60,000 cells/mm3;
   * Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve the required hemoglobin is permitted).

   2.5 Serum creatinine < 3 mg/dL (265 μmol/L) within 2 weeks prior to registration; 2.6 Total bilirubin < 2.5 mg/dL (43 μmol/L) within 2 weeks prior to registration; 2.7 Pregnancy test (urine dipstick or serum) for women of childbearing potential within 2 weeks prior to registration;
3. ≥ 18 years of age;
4. Zubrod performance status 0-2 for patients with breast or prostate primaries; Zubrod performance status 0-1 for patients with lung primaries;
5. Patients receiving systemic chemotherapy or hormonal therapy are eligible for this study. See Sections 6.0 and 7.0 for further details. Note: All patients must complete external beam radiation therapy ≥ 14 days prior to registration. If patients have undergone CyberKnife treatment, treatment must be completed ≥ 14 days prior to registration.
6. Patients may have received prior oral bisphosphonate therapy, such as Fosamax® or similar medications. Duration of bisphosphonate treatment prior to study entry must be documented, and all bisphosphonates other than the study drug must be discontinued prior to registration.
7. Women of childbearing potential and male participants must agree to practice an adequate means of birth control throughout their participation in the study.
8. Patient must sign study specific informed consent prior to study entry.

Exclusion Criteria

1. Patients with brain metastases and/or spinal cord compression are excluded. Note: Patients with no evidence of disease in the brain after treatment for brain metastases are eligible.
2. Patients with painful bone metastases are not permitted until these bone metastases are successfully treated (for example by external beam irradiation) prior to registration, and the patient has stable pain for at least 2 weeks after that treatment (Stable pain is defined for this study as a patient response of 1, 2, or 3 on Questions 4 and 5 of The Brief Pain Inventory (BPI).
3. Prior treatment with Strontium-89 or Samarium-153 for bone metastases.
4. Treatment for more than 6 months with IV bisphosphonates prior to study entry;
5. Treatment with calcitonin, mithramycin, or gallium nitrate within 2 weeks prior to registration
6. Severe, active co-morbidity, defined as follows:

   6.1 Evidence in the six months prior to study entry of uncontrolled congestive heart failure, hypertension refractory to treatment, or symptomatic coronary artery disease; 6.2 Current, active dental problems within 4 weeks of registration, including infection of the teeth or jawbone (maxilla or mandible); dental or fixture trauma; current or prior diagnosis of osteonecrosis of the jaw (ONJ); exposed bone in the mouth; or slow healing after dental procedures; 6.3 Dental surgery (e.g., extractions, implants) within 6 weeks of study entry and while receiving study treatment; for patients who require dental surgery, there are no data to suggest whether discontinuation of bisphosphonate treatment reduces the risk of osteonecrosis of the jaw (ONJ) [see Section 7.2.4].

   6.4 Acquired Immune Deficiency Syndrome (AIDS) based upon current Center for Disease Control (CDC) definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immuno-compromised patients.
7. Pregnant or lactating patients are excluded, as treatment may be harmful to embryos and/or nursing infants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2006-07-11 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2017-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Seider, MD, PhD, FACR, Study Chair — Summa Center for Cancer Care at Akron City Hospital
Locations (147):
- United States (147):
  - Providence Cancer Center at Providence Hospital, Mobile, Alabama
  - Roy and Patricia Disney Family Cancer Center at Providence Saint Joseph Medical Center, Burbank, California
  - Mercy Cancer Center at Mercy San Juan Medical Center, Carmichael, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Robert and Beverly Lewis Family Cancer Care Center at Pomona Valley Hospital Medical Center, Pomona, California
  - Radiation Oncology Center - Roseville, Roseville, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - General Robert Huyser Cancer Center at David Grant Medical Center, Travis Air Force Base, California
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Integrated Community Oncology Network at Southside Cancer Center, Jacksonville, Florida
  - Baptist Medical Center South, Jacksonville, Florida
  - Integrated Community Oncology Network, Jacksonville Beach, Florida
  - Miami Cancer Center at Mercy Hospital, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Integrated Community Oncology Network - Orange Park, Orange Park, Florida
  - Florida Cancer Center - Palatka, Palatka, Florida
  - Bay Medical, Panama City, Florida
  - Flagler Cancer Center, Saint Augustine, Florida
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - John B. Amos Cancer Center, Columbus, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Good Samaritan Cancer Care Center at Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Veterans Affairs Medical Center - Hines, Hines, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Advocate Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Cancer Institute at St. John's Hospital, Springfield, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Center for Cancer Care at Goshen General Hospital, Goshen, Indiana
  - Cancer Center at Ball Memorial Hospital, Muncie, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Central Baptist Hospital, Lexington, Kentucky
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - Central Maine Comprehensive Cancer Center at Central Maine Medical Center, Lewiston, Maine
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - Hudner Oncology Center at Saint Anne's Hospital - Fall River, Fall River, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Princeton Radiation Oncology Center, Jamesburg, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - University Medical Center at Princeton, Princeton, New Jersey
  - Franklin & Edith Scarpa Regional Cancer Center at South Jersey Healthcare, Vineland, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - New Mexico Cancer Center, Albuquerque, New Mexico
  - New York Methodist Hospital, Brooklyn, New York
  - Sands Cancer Center, Canandaigua, New York
  - Fitzpatrick Cancer Center at Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - Highland Hospital of Rochester, Rochester, New York
  - Lipson Cancer and Blood Center at Rochester General Hospital, Rochester, New York
  - University Radiation Oncology at Parkridge Hospital, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Trinity CancerCare Center, Minot, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Radiation Oncology Center, Alliance, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Mercy Cancer Center at Mercy Medical Center, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - MedCentral - Mansfield Hospital, Mansfield, Ohio
  - Cancer Care Center, Incorporated, Salem, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson Air Force Base, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - UPMC Cancer Center at Beaver Medical Center, Beaver, Pennsylvania
  - UPMC Cancer Center at Jefferson Regional Medical Center, Clairton, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - UPMC Cancer Center - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Cancer Center at the John P. Murtha Pavilion, Johnstown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC - Moon, Moon Township, Pennsylvania
  - UPMC Cancer Center - Natrona Heights, Natrona Heights, Pennsylvania
  - Jameson Memorial Hospital - North Campus, New Castle, Pennsylvania
  - UPMC - Shadyside, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Presbyterian, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC St. Margaret, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Passavant, Pittsburgh, Pennsylvania
  - UPMC Cancer Center - Upper St. Clair, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - UPMC Cancer Center - Uniontown, Uniontown, Pennsylvania
  - Washington Hospital Cancer Center, Washington, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - St. Francis Hospital, Federal Way, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Theda Care Cancer Institute, Appleton, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Riverview UW Cancer Center at Riverview Hospital, Wisconsin Rapids, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Seider MJ, Pugh SL, Langer C, Wyatt G, Demas W, Rashtian A, Clausen CL, Derdel JD, Cleary SF, Peters CA, Ramalingam A, Clarkson JE, Tomblyn M, Rabinovitch RA, Kachnic LA, Berk LB; NRG Oncology. Randomized phase III trial to evaluate radiopharmaceuticals and zoledronic acid in the palliation of osteoblastic metastases from lung, breast, and prostate cancer: report of the NRG Oncology RTOG 0517 trial. Ann Nucl Med. 2018 Oct;32(8):553-560. doi: 10.1007/s12149-018-1278-4. Epub 2018 Aug 9. PMID 30094545
- Available data/document: Individual Participant Data Set: NCT00365105 — https://nctn-data-archive.nci.nih.gov/ — Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zoledronic Acid | Zoledronic Acid + Radiopharmaceuticals
Started | 129 | 132
Eligible | 124 | 124
Eligible With Adverse Event Data | 123 | 124
Completed (Subjects contributing any data to analysis are considered to have completed the study) | 124 | 124
Not Completed | 5 | 8
Not completed — Protocol Violation | 5 | 8

BASELINE CHARACTERISTICS:
Population: Eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid | Zoledronic Acid + Radiopharmaceuticals | Total
Number analyzed (Participants) | 124 | 124 | 248
Age, Continuous [Median (Full Range); unit: years] | 68 [25 to 88] | 68 [32 to 90] | 68 [25 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 48 | 95
  Male | 77 | 76 | 153

OUTCOME MEASURES:

1. Primary Outcome: Time to Development of a Malignant Skeletal-related Events (SRE)
Description: Median time to development of a malignant skeletal related event (SRE), which is defined as a pathological bone fracture, spinal cord compression, surgery to bone or radiation to bone is estimated using Kaplan-Meier method. The time of failure was measured from date of randomization to the date of a documented SRE. The analysis was planned to occur after 257 SRE have been observed, unless the criteria for early stopping are met.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 80.1 months.
Population: Eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Zoledronic Acid | Zoledronic Acid + Radiopharmaceuticals
Number analyzed (Participants) | 124 | 124
months | 29.9 [25.8 to 37.4] | 27.4 [21.2 to 35.34]
Statistical Analysis 1: Comparison: Zoledronic Acid vs Zoledronic Acid + Radiopharmaceuticals; Assuming an exponential distribution, the weighted yearly SRE hazard rate for patients treated with bisphosphonates only is 0.7991 which translates to a median time to SRE of 10.4 months. The study was designed to show a 33% relative reduction in the yearly SRE hazard rate, i.e. 15.6 months median time to SRE. Using a two-sided log-rank test assuming a type I error of 0.05, one planned interim analysis with 90% statistical power, 257 SREs are required with a total of 316 patients; Test type: Superiority or Other; p = 0.844, Log Rank; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.70 to 1.54]

2. Secondary Outcome: Number of Patients Experiencing a Skeletal-related Event (SRE) Within One Year
Description: Skeletal-related events are defined as a pathological bone fracture, spinal cord compression, surgery to bone or radiation to bone.
Time Frame: From randomization to 1 year
Population: Eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Zoledronic Acid | Zoledronic Acid + Radiopharmaceuticals
Number analyzed (Participants) | 124 | 124
Participants | 28 | 20
Statistical Analysis 1: Comparison: Zoledronic Acid vs Zoledronic Acid + Radiopharmaceuticals; Test type: Superiority — The power of detecting an improvement from 55% in the control arm to 41% in the experimental arm with a two-sided Fisher's exact test at alpha 0.05 is 66%; p = 0.26, Fisher Exact

3. Secondary Outcome: Overall Survival
Description: Overall survival time is defined as time from randomization to the date of death from any cause. Overall survival rates are estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 101.7 months.
Population: Eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Zoledronic Acid | Zoledronic Acid + Radiopharmaceuticals
Number analyzed (Participants) | 124 | 124
months | 32.1 [22.1 to 37.5] | 26.9 [20.4 to 33.6]
Statistical Analysis 1: Comparison: Zoledronic Acid vs Zoledronic Acid + Radiopharmaceuticals; Assuming the disease site distribution is 40%, 40%, and 20% from prostate, breast, and lung cancer populations, respectively, the weighted yearly death rate for patients treated with bisphosphonates only is 0.4390, translating to a median overall survival time of 18.9 months assuming an exponential distribution. Statistical power to detect a relative difference of 33% in the yearly death rate is 70% using a two-sided log-rank test at a 0.05 significance level and 87% to detect 50% difference; Test type: Superiority; p = 0.37, Log Rank; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.86 to 1.52]

4. Secondary Outcome: Change in Functional Assessment of Cancer Therapy - General (FACT-G) at One Year
Description: The FACT-G is a validated 27-item measure in which a higher score represents higher quality of life (QOL). Physical, functional, social and emotional well-being subscale scores are added together to form the FACT-G total score. Responses range from 0=Not a lot to 4=Very much. Certain items must be reversed before being added, by subtracting the response from 4. Subscale items are added together, multiplied by the number of items in the subscale, then divided by the number of items answered to obtain subscale totals. Total score ranges from 0-108; physical, social and functional subscales from 0-28; emotional subscale from 0-24. Each subscale requires at least 50% of the items to be completed while the overall response rate must be greater than 80%. If items are missing the subscale scores can be prorated. Change score at one year is calculated as one year score - baseline score with a positive change score indicating improvement in QOL.
Time Frame: Baseline and 1 year
Population: Eligible patients with FACT-G scores at baseline and one year
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Zoledronic Acid | Zoledronic Acid + Radiopharmaceuticals
Number analyzed (Participants) | 62 | 59
units on a scale
  FACT-G Total: number analyzed (Participants) | 62 | 55
  FACT-G Total | -1 [-8 to 5] | -2 [-11 to 4]
  Physical Well-Being: number analyzed (Participants) | 62 | 58
  Physical Well-Being | -1 [-4 to 1] | -1 [-4 to 2]
  Social/Family Well-Being: number analyzed (Participants) | 62 | 58
  Social/Family Well-Being | 0 [-1 to 2] | 0 [-2 to 2]
  Emotional Well-Being: number analyzed (Participants) | 62 | 57
  Emotional Well-Being | 0 [-1 to 3] | 0 [-2 to 2]
  Functional Well-Being: number analyzed (Participants) | 62 | 57
  Functional Well-Being | 0 [-4 to 2] | 0 [-4 to 1]
Statistical Analysis 1: Comparison: Zoledronic Acid vs Zoledronic Acid + Radiopharmaceuticals; FACT-G Total; Test type: Superiority; p = 0.96, Wilcoxon (Mann-Whitney) — Two-sided significance level of 0.01
Statistical Analysis 2: Comparison: Zoledronic Acid vs Zoledronic Acid + Radiopharmaceuticals; Physical Well-Being; Test type: Superiority; p = 0.97, Wilcoxon (Mann-Whitney) — Two-sided significance level of 0.01
Statistical Analysis 3: Comparison: Zoledronic Acid vs Zoledronic Acid + Radiopharmaceuticals; Social/Family Well-Being; Test type: Superiority; p = 0.57, Wilcoxon (Mann-Whitney) — Two-sided significance level of 0.01
Statistical Analysis 4: Comparison: Zoledronic Acid vs Zoledronic Acid + Radiopharmaceuticals; Emotional Well-Being; Test type: Superiority; p = 0.70, Wilcoxon (Mann-Whitney) — Two-sided significance level of 0.01
Statistical Analysis 5: Comparison: Zoledronic Acid vs Zoledronic Acid + Radiopharmaceuticals; Functional Well-Being; Test type: Superiority; p = 0.46, Wilcoxon (Mann-Whitney) — Two-sided significance level of 0.01

5. Secondary Outcome: Change in Brief Pain Inventory (BPI) at One Year
Description: The Brief Pain Inventory (BPI) is a measurement tool for assessing clinical pain. The BPI assesses severity (pain at its "worst," "least," "average," and "now"), and interference (how much pain has interfered with seven daily activities, including general activity, walking, work, mood, enjoyment of life, relations with others, and sleep). Patients rate the severity of their pain and the degree to which their pain interferes with common dimensions of feeling and function on a scale of 0 to 10, with 0=no pain/interference and 10=interferes completely/worst pain imaginable.
Time Frame: Baseline and 1 year
Population: Eligible patients with baseline and one-year BPI score
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Zoledronic Acid | Zoledronic Acid + Radiopharmaceuticals
Number analyzed (Participants) | 54 | 51
units on a scale | 1 [-5 to 9] | 0 [-6 to 7]
Statistical Analysis 1: Comparison: Zoledronic Acid vs Zoledronic Acid + Radiopharmaceuticals; Test type: Superiority; p = 0.99, Wilcoxon (Mann-Whitney) — 2-sided significance level of 0.05

6. Secondary Outcome: Change in EuroQol-5 Dimension 3-level (EQ-5D-3L) at One Year
Description: The EQ-5D-3L is a 2-part self-assessment questionnaire. First part is 5 items (mobility, self care, usual activities, pain/discomfort, anxiety/depression) each with 3 problem levels (1-none, 2-moderate, 3-extreme). The 5-item index score is transformed into a utility score between 0 (worst health state) and 1 (best health state). The 2nd part is a visual analogue scale (VAS) valuing current health state, measured on a 20-cm 10-point interval scale. Worst imaginable health state is scored as 0 at the bottom of the scale, and best imaginable health state is scored as 100 at the top. Change at one year is calculated as one-year score - baseline score with positive change indicating improved quality of life.
Time Frame: Baseline and 1 year
Population: Eligible patients with EQ-5D-3L scores at baseline and one year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zoledronic Acid | Zoledronic Acid + Radiopharmaceuticals
Number analyzed (Participants) | 53 | 51
units on a scale
  Index Score | -0.04 (0.14) | -0.06 (0.15)
  VAS Score: number analyzed (Participants) | 50 | 44
  VAS Score | -1.20 (20.43) | -6.70 (15.70)
Statistical Analysis 1: Comparison: Zoledronic Acid vs Zoledronic Acid + Radiopharmaceuticals; Index Score; Test type: Superiority; p = 0.43, t-test, 2 sided — Significance level of 0.05
Statistical Analysis 2: Comparison: Zoledronic Acid vs Zoledronic Acid + Radiopharmaceuticals; VAS Score; Test type: Superiority; p = 0.15, t-test, 2 sided — Significance level of 0.05

ADVERSE EVENTS:
Description: Eligible patients with adverse event data. Patients experiencing more than one of a given adverse event are counted only once for that adverse event.
Arm/Group | Zoledronic Acid | Zoledronic Acid + Radiopharmaceuticals
Serious Adverse Events (participants affected / at risk) | 31/123 | 37/124
Other Adverse Events (participants affected / at risk) | 102/123 | 108/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid (N=123) | Zoledronic Acid + Radiopharmaceuticals (N=124)
Blood/bone marrow - Other: (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Hemoglobin (Blood and lymphatic system disorders) | 6 | 10
Atrial fibrillation (Cardiac disorders) | 1 | 2
Cardiac General - Other: (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Sick Sinus Syndrome (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 2
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Diplopia (Eye disorders) | 1 | 0
Abdominal pain NOS (Gastrointestinal disorders) | 2 | 1
Colonic obstruction (Gastrointestinal disorders) | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea NOS (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal - Other: (Gastrointestinal disorders) | 0 | 1
Ileal haemorrhage (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal stricture NOS (Gastrointestinal disorders) | 0 | 1
Vomiting NOS (Gastrointestinal disorders) | 2 | 2
Chest pain (General disorders) | 2 | 0
Death NOS (General disorders) | 1 | 1
Disease progression NOS (General disorders) | 3 | 2
Edema: limb: (General disorders) | 1 | 0
Fatigue (General disorders) | 4 | 0
Gait abnormal NOS (General disorders) | 1 | 0
Pain NOS (General disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 1 | 0
Bladder infection NOS (Infections and infestations) | 1 | 1
Bone infection NOS (Infections and infestations) | 1 | 0
Bronchitis NOS (Infections and infestations) | 1 | 0
Infection - Other: (Infections and infestations) | 0 | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Bladder (urinary) (Infections and infestations) | 0 | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Catheter-related (Infections and infestations) | 1 | 0
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Lung (pneumonia) (Infections and infestations) | 1 | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Pleura (empyema) (Infections and infestations) | 0 | 1
Infection with unknown ANC: Urinary tract NOS (Infections and infestations) | 1 | 1
Pneumonia NOS (Infections and infestations) | 2 | 2
Sepsis NOS (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Fracture NOS (Injury, poisoning and procedural complications) | 2 | 3
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 1
Blood creatinine increased (Investigations) | 4 | 3
Leukopenia NOS (Investigations) | 2 | 1
Lymphopenia (Investigations) | 0 | 1
Metabolic/laboratory - Other: (Investigations) | 1 | 0
Neutrophil count (Investigations) | 2 | 2
Platelet count decreased (Investigations) | 1 | 7
Prothrombin time prolonged (Investigations) | 1 | 1
Troponin T increased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 2 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 2
Osteoporosis NOS (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Ataxia (Nervous system disorders) | 2 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 2
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 1 | 0
Neurology - Other: (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 0
Syncope vasovagal (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 1
Bladder obstruction (Renal and urinary disorders) | 0 | 1
Renal failure NOS (Renal and urinary disorders) | 2 | 1
Renal/genitourinary - Other: (Renal and urinary disorders) | 1 | 1
Urethral obstruction (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Pulmonary/upper respiratory - Other: (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Ulceration: (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension NOS (Vascular disorders) | 5 | 2
Thrombosis (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid (N=123) | Zoledronic Acid + Radiopharmaceuticals (N=124)
Hemoglobin (Blood and lymphatic system disorders) | 56 | 73
Ocular/visual - Other: (Eye disorders) | 6 | 3
Abdominal pain NOS (Gastrointestinal disorders) | 8 | 9
Constipation (Gastrointestinal disorders) | 29 | 26
Diarrhoea NOS (Gastrointestinal disorders) | 19 | 18
Dry mouth (Gastrointestinal disorders) | 2 | 6
Dyspepsia (Gastrointestinal disorders) | 7 | 3
Nausea (Gastrointestinal disorders) | 30 | 31
Stomatitis (Gastrointestinal disorders) | 7 | 9
Vomiting NOS (Gastrointestinal disorders) | 12 | 19
Chest pain (General disorders) | 11 | 2
Disease progression NOS (General disorders) | 4 | 6
Edema: limb: (General disorders) | 28 | 25
Fatigue (General disorders) | 68 | 77
Pain - Other: (General disorders) | 13 | 8
Pain NOS (General disorders) | 10 | 4
Pyrexia (General disorders) | 5 | 7
Pneumonia NOS (Infections and infestations) | 1 | 6
Respiratory tract infection NOS (Infections and infestations) | 1 | 6
Ecchymosis (Injury, poisoning and procedural complications) | 2 | 7
Fracture NOS (Injury, poisoning and procedural complications) | 6 | 4
Alanine aminotransferase increased (Investigations) | 12 | 14
Aspartate aminotransferase increased (Investigations) | 23 | 21
Blood alkaline phosphatase increased (Investigations) | 31 | 27
Blood bilirubin increased (Investigations) | 7 | 5
Blood creatinine increased (Investigations) | 31 | 28
Leukopenia NOS (Investigations) | 26 | 42
Lymphopenia (Investigations) | 13 | 13
Neutrophil count (Investigations) | 15 | 32
Platelet count decreased (Investigations) | 19 | 52
Weight decreased (Investigations) | 16 | 22
Weight increased (Investigations) | 2 | 8
Anorexia (Metabolism and nutrition disorders) | 23 | 29
Dehydration (Metabolism and nutrition disorders) | 8 | 5
Hypercalcaemia (Metabolism and nutrition disorders) | 10 | 4
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 38 | 32
Hyperkalaemia (Metabolism and nutrition disorders) | 10 | 9
Hypoalbuminemia (Metabolism and nutrition disorders) | 26 | 20
Hypocalcemia (Metabolism and nutrition disorders) | 17 | 26
Hypokalemia (Metabolism and nutrition disorders) | 8 | 13
Hyponatremia (Metabolism and nutrition disorders) | 16 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 | 29
Arthritis NOS (Musculoskeletal and connective tissue disorders) | 6 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 39 | 37
Bone pain (Musculoskeletal and connective tissue disorders) | 40 | 46
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 9 | 10
Muscle weakness, generalized or specific area (not due to neuropathy): Extremity-lower (Musculoskeletal and connective tissue disorders) | 6 | 7
Musculoskeletal/soft tissue - Other: (Musculoskeletal and connective tissue disorders) | 3 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 12
Neck pain (Musculoskeletal and connective tissue disorders) | 9 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 | 20
Dizziness (Nervous system disorders) | 21 | 18
Dysgeusia (Nervous system disorders) | 8 | 3
Headache (Nervous system disorders) | 15 | 14
Peripheral motor neuropathy (Nervous system disorders) | 7 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 23 | 18
Anxiety (Psychiatric disorders) | 6 | 9
Depression (Psychiatric disorders) | 11 | 12
Insomnia (Psychiatric disorders) | 12 | 19
Pollakiuria (Renal and urinary disorders) | 9 | 14
Renal/genitourinary - Other: (Renal and urinary disorders) | 4 | 6
Urinary incontinence (Renal and urinary disorders) | 8 | 6
Urinary retention (Renal and urinary disorders) | 5 | 7
Pelvic pain NOS (Reproductive system and breast disorders) | 8 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 | 32
Pulmonary/upper respiratory - Other: (Respiratory, thoracic and mediastinal disorders) | 4 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 12
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 7 | 2
Dermatology/skin - Other: (Skin and subcutaneous tissue disorders) | 9 | 6
Localised exfoliation (Skin and subcutaneous tissue disorders) | 4 | 6
Hot flushes NOS (Vascular disorders) | 16 | 17
Hypertension NOS (Vascular disorders) | 6 | 4
Hypotension NOS (Vascular disorders) | 4 | 7

LIMITATIONS AND CAVEATS:
This study stopped accrual early with 261 accrued out of 352 planned, due to a lower than expected rate of skeletal related events in the control arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.